CLINICAL TRIAL: NCT02995668
Title: Influencia de un Entrenamiento Preoperatorio de propiocepción y Equilibrio en Pacientes Con Artrosis Severa de Rodilla en Espera Para la intervención de Artroplastia Total
Brief Title: Effects of Specific Balance Training Prior TKR Surgery in the Early Postoperative Outcomes
Acronym: PRE_TKR_BLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Jose María Blasco Igual, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRE_ATR_BALANCE
Record Dates: First submitted 2016-12-11; First posted 2016-12-16 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis; Aging
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Non-active comparator
- Strength-Function (Active Comparator): Active comparator
  Interventions: Other: Strength-Function
- Balance-Proprioception (Experimental): Experimental
  Interventions: Other: Strength-Function; Other: Balance-Proprioception

INTERVENTIONS:
Other: Strength-Function — Preoperative functional and strength capabilities training.
  Arms: Balance-Proprioception; Strength-Function
Other: Balance-Proprioception — Preoperative proprioceptive and balance capabilities training
  Arms: Balance-Proprioception

SUMMARY:
Knee osteoarthritis is one of the most common pathologies in old people, and the leading cause of pain and disability. Symptoms include joint pain, stiffness, limited mobility, functional impairment and proprioceptive deficit. When conservative treatments fail to control these symptoms, a total knee replacement (TKR) is the chosen treatment, mainly because of its efficacy on pain relief. In recent decades, this surgical procedure has been soared, and it has also aroused the interest of researches about the patients' outcomes after surgery.

Despite the TKR results in good reported outcomes, after surgery patients may manifest persistent pain and problems affecting to their functionality, stability, walking speed, proprioception, motor control, risk of falling and therefore to their quality of life. In more than a third of the cases, those deficiencies may be extended after surgery from six months to one year, when subjects use to achieve the plateau functional values.

Traditional rehabilitation programs have been usually focused on improving muscle strength of the lower limbs as well as the functionality with specific exercises to achieve this purpose, and to a lesser extent on balance and proprioception exercises. Evidence supports this approach. Yet, task-oriented rehabilitation focusing on balance enhancement may be one of the most important factors for a complete rehabilitation, since benefits of proprioceptive and balance trainings may range from better stability and motor control, improvements in both static and dynamic balance and enhanced functionality. Indeed, recent studies have shown that the combination of traditional functional rehabilitation together with balance training may help to restore functional deficits to a larger extent than usual therapy, and based on a systematic review published (Moutzori, 2015) and in our previous works (Roig, 2016), sensori-motor training is an acceptable adjust to usual physiotherapy care .

Looking into the effect of preoperative trainings or education before TKR surgery, it is aimed at improving the physical function, but also managing the expectations of the surgery for a better recovery. There is from low to moderate evidence about the effects of TKR pre-interventional training programs, and some authors have argued that the effects are too small to be consider clinically relevant.

In general, the preoperative program is usually focused on functional and strengthening exercises. Despite of proprioception is used in the clinical practice for the prevention and recovery of many orthopedics injuries, the amount of evidence about the effects of proprioceptive training programs for knee and hip replacement is not large, few works compares pre-habilitation and post-rehabilitation programs, and there is not systematically reviewed evidence reporting the efficacy of balance and proprioceptive pre-interventional training programs.

In this framework, this aimed at evaluating the effects of specific-task oriented proprioceptive and balance training programs when conducted by patients undergoing TKR before and after surgery, and will compare these effects to the outcomes achieved with traditional strength-functional programs, as well as to no specific prehabilitation training.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 and 80.
* Subjects with severe knee osteoarthritis that have not been operated before.
* Patients will be operated with the same total replacement prosthesis and same surgical procedure.
* The score in Berg scale must be greater than 21, indicating a medium-low risk of falling.
* The score of the Mini-Mental State Examination must be equal or greater than 20, which means they do not have moderate or severe cognitive impairment.
* Once the informed consent is read and explained, patients must accept and agree to participate in the study.

Exclusion Criteria:

* Patient with morphological alterations hip or ankle (also knee).
* Patient with suspected deep vein thrombosis or post-surgical infection of the operated knee.
* Patient with pathology of central origin (i.e. cerebellar) that could interfere with the results of the test of balance or strength
* Patient with vestibular pathology that could interfere with the results of the test of balance

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  http://www.koos.nu/KOOSusersguide2012.pdf
Berg Balance Scale (BBS) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Overall state of balance. Balance among older people with impairment in balance function by assessing the performance of functional tasks from the total score achieved in the 14 items test

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Dynamic balance assessment. Also points at the risk of falling. Time of getting up from a chair, walk three meters, come back and sit again, measured in seconds
Knee Range of Mobility (ROM) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Knee Range of Mobility (Flexion, Extension) in degrees
Quadriceps Strength | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Electronic dynamometer in Newton
Euro Quality of Life 5 Dimension (Euro-QoL-5D) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Quality of Life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Blasco, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dominguez-Navarro F, Silvestre-Munoz A, Igual-Camacho C, Diaz-Diaz B, Torrella JV, Rodrigo J, Paya-Rubio A, Roig-Casasus S, Blasco JM. A randomized controlled trial assessing the effects of preoperative strengthening plus balance training on balance and functional outcome up to 1 year following total knee replacement. Knee Surg Sports Traumatol Arthrosc. 2021 Mar;29(3):838-848. doi: 10.1007/s00167-020-06029-x. Epub 2020 Apr 27. PMID 32342139